CLINICAL TRIAL: NCT01918579
Title: Efficacy of Point-of-care (POC) C-reactive Protein Testing to Reduce Inappropriate Use of Antibiotics for Acute Respiratory Infections (ARIs) in the Primary Health Care Setting of Hanoi - a Randomized Controlled Trial
Brief Title: C Reactive Protein (CRP) Intervention to Reduce Inappropriate Antibiotic Prescriptions in the Primary Healthcare Setting
Acronym: CRP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oxford University Clinical Research Unit, Vietnam (Other)
Collaborators: National Hospital for Tropical Diseases, Hanoi, Vietnam (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 05HN
Record Dates: First submitted 2013-08-06; First posted 2013-08-07 (Estimated); Last update posted 2016-11-15 (Estimated); Status verified 2014-06

CONDITIONS: Acute Respiratory Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- CRP intervention (Experimental): Patients will be tested by rapid POC CRP test
  Interventions: Procedure: Patients will be tested by rapid POC CRP test
- Control (No Intervention): Patients will not be tested by rapid POC CRP test

INTERVENTIONS:
Procedure: Patients will be tested by rapid POC CRP test — Patient will be tested with CRP test. Treatment decisions including any antibiotics prescribed will be based on test results and clinical judgement. Treatment choices are not recommended/prescribed by the study protocol.
  Arms: CRP intervention

SUMMARY:
Many studies have showed that rapid point-of-care (POC) c-reactive protein (CRP) test can reduce inappropriate use of antibiotic at primary health care level. In Vietnam, prevalence of antibiotic abuse for community acute respiratory infection has been reported. This study will test the hypothesis that CRP POC testing for patients with non-severe acute respiratory illness at primary healthcare stations reduces inappropriate antibiotic use safely.

The study will be conducted at ten district health care facilities in Hanoi, Viet Nam. Investigators intend to enroll 2,000 participants aged 6-65 years with non-severe acute respiratory infection. Patients will be randomly allocated to the control or the intervention arm. Participants in the control group will be treated according to routine care. Participants in the intervention arm will have a CRP test, the results of which will be available to the health care practitioner to contribute to their diagnosis and treatment decisions.

All patients will be followed-up via telephone call after 14 days. The study will compare the proportion of patients in each arm receiving any antibiotics within 2 weeks of study enrollment.

ELIGIBILITY:
Inclusion Criteria:

* Patients, aged 6 to 65 years, that visit one of the 10 selected primary healthcare centers
* Suspected to have acute respiratory tract infection (ARI) by treating physician
* Informed consent

Exclusion Criteria:

* Severe respiratory disease as determined by treating doctor
* Any disease or symptom requiring hospital referral as determined by treating doctor
* Immunosuppressed patients (e.g. HIV, long term steroid use)
* Suspicion of tuberculosis
* Evidence of acute or chronic liver disease (e.g. hepatitis or cirrhosis due to any cause)
* Past medical history of: neoplastic disease, congestive cardiac failure, chronic obstructive pulmonary disease, insulin-dependent diabetes or renal disease
* Pregnancy
* No access to telephone
* Not able to come for follow up visit on day 3 or 4.
* Already taking antibiotics at the time of presentation
* Symptoms present for more than 2 weeks
* Presence of any sign of severe diseases as defined by the British Thoracic Society modified CRP-65 system for severity scoring of pneumonia in primary care.

For children (Age ≥ 6 years and < 16 years) additional exclusion criteria include: Tachypnea, signs of chest wall in drawing, reduced consciousness, confusion, dehydration, hypothermia, severe malnutrition, unable to feed or drink, vomiting, and convulsions.

Ages: 6 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 2037 (Actual)
Dates: Start 2014-03; Primary Completion 2015-07 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Proportion of patients receiving any antibiotic | 2 weeks
  Number of patients receiving any antibiotic within 2 weeks of study enrollment as a proportion of the total number of patients.

SECONDARY OUTCOMES:
Duration of symptoms | 2 weeks
  Number of days that symptoms (including fever or any respiratory symptom) endure.
Frequency of re-consultation | 2 weeks
  Number of visits to a health care practitioner during the 14 day follow-up.
Frequency of serious adverse events | 2 weeks
  Number of serious adverse events which occur during the 14 day follow-up period.

OTHER OUTCOMES:
The attitudes and satisfaction of patients and health center staff towards the test. | 2 weeks
  Patients and health center staff will be interviewed by structured questionnaire to assess their attitudes and satisfaction toward the intervention.
  The Likert scale will be used for quantifying attitude orientation of interviewees

CONTACTS AND LOCATIONS:
Overall Officials: Heiman FL Wertheim, M.D,Ph.D, Study Director — Oxford University Clinical Research Unit
Locations (1):
- National Hospital for Tropical Diseases, Hanoi, Hanoi, Vietnam

REFERENCES:
- [Derived] Haenssgen MJ, Charoenboon N, Do NTT, Althaus T, Khine Zaw Y, Wertheim HFL, Lubell Y. How context can impact clinical trials: a multi-country qualitative case study comparison of diagnostic biomarker test interventions. Trials. 2019 Feb 8;20(1):111. doi: 10.1186/s13063-019-3215-9. PMID 30736818
- [Derived] Do NT, Ta NT, Tran NT, Than HM, Vu BT, Hoang LB, van Doorn HR, Vu DT, Cals JW, Chandna A, Lubell Y, Nadjm B, Thwaites G, Wolbers M, Nguyen KV, Wertheim HF. Point-of-care C-reactive protein testing to reduce inappropriate use of antibiotics for non-severe acute respiratory infections in Vietnamese primary health care: a randomised controlled trial. Lancet Glob Health. 2016 Sep;4(9):e633-41. doi: 10.1016/S2214-109X(16)30142-5. Epub 2016 Aug 3. PMID 27495137
- See also: Oxford University Clinical Research Unit, Viet Nam — http://www.oucru.org